CLINICAL TRIAL: NCT03434457
Title: Maternal Adversity, Vulnerability and Neurodevelopment
Acronym: MAVAN
Status: Completed | Type: Observational
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The JPB Foundation (Unknown); Ludmer Family Foundation (Unknown); Norlien Foundation (Other); WOCO Foundation (Unknown); Blema & Arnold Steinberg Family Foundation (Unknown); McGill University (Other); Jacobs Foundation (Unknown)
Responsible Party: Principal Investigator, Michael J Meaney, James McGill professor, Douglas Mental Health University Institute
Other Study IDs: DouglasMHU
Record Dates: First submitted 2018-01-30; First posted 2018-02-15 (Actual); Results first posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse); Infant Development; Infant Behavior
Keywords: Fetal growth retardation; Early adversity; Depressive Symptoms
MeSH Terms: conditions — Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders; Infant Behavior; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prenatal and 3 to 72 months

SUMMARY:
Maternal Adversity Vulnerability and Neurodevelopment (MAVAN) project is a prospective community-based, pregnancy and birth cohort of Canadian mother-child dyads. The main objective of MAVAN project is to examine the pre- and postnatal influences, and their interaction, in determining individual differences in children development. The MAVAN project is designed to examine the consequences of fetal adversity as a function of the quality of the postnatal environment, focusing on mother-infant interactions.

DETAILED DESCRIPTION:
In 2003 the Canadian Institutes of Health Research (CIHR) funded an ambitious and internationally unique study on the development of individual differences in vulnerability for mental illness. Increasing evidence indicates that many forms of mental illness as well as diabetes and cardiovascular disease are best considered as developmental disorders where vulnerability emerges as a function of genetic and epigenetic events. Frank pathology then develops as a function of the continuous interaction between underlying vulnerability and prevailing environmental triggers. The critical question is that of understanding the mechanisms by which specific forms of gene x environment interactions in perinatal life define the level of vulnerability/resistance to illness.

Maternal adversity during fetal life including maternal stress (as well as depression), low social support, poor maternal nutrition, and tobacco/alcohol consumption predict both preterm labour and intrauterine growth restriction. These birth outcomes, in turn, represent major epidemiological risk factors for heart disease, diabetes, and depression in adulthood, and neurodevelopmental impairments in children. Postnatal maternal adversity compromises maternal care/behaviour and infant development, and predicts increased risk for obesity, heart disease, attentional deficit disorders (ADD), drug abuse, and depression. Despite the enormous potential for the interaction of prenatal and postnatal influences, research has largely been restricted to the effects of events occurring during only one developmental period which, among other things, ignores the potential importance of 'protective' factors operating at later stages in life. Moreover, the underlying mechanisms by which perinatal adversity might directly affect neurocognitive development have been very poorly studied.

The investigators proposed an innovative research program that focuses on child development using a longitudinal, within-subject design examining neural and cognitive/emotional outcomes as a function of genomic and epigenomic factors. These studies focus on 500 mother-infant dyads drawn from two human studies (Montreal & Hamilton). Assessment of maternal wellbeing and infant development (cognition, socio-emotional development, temperament, and brain structure) trajectories are undertaken from mid-pregnancy until 10 years of age. Genomic and epigenomic approaches were used to assess genetic vulnerability in these populations using a GWAS approach. This represents the first longitudinal study linking neurocognitive/behavioural function with structural neurodevelopment through neuroimaging and genetic vulnerability in humans, in the presence or absence of maternal adversity. The ability to identify postnatal events that serve to reverse a condition of vulnerability has enormous implications for the development of prevention /intervention programs reducing the future rates of a broad spectrum of chronic illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women recruited when they attending antenatal care clinics at the time of routine ultrasound or through advertisements at hospitals (usually at 13 to 20 weeks' gestation). Women were included in the study if they were 18 years of age or older, and fluent in either English or French. Only babies born at 37 weeks or later and above 2000 g were included in the MAVAN cohort.

Exclusion Criteria:

* Exclusion criteria included serious obstetric complications during the pregnancy or delivery of the child, extremely low birth weight, prematurity (less than 37 weeks of gestation), or any congenital diseases.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Our community sample consisted of mothers recruited in Montréal (Québec) and Hamilton (Ontario), Canada, at 13 to 20 weeks' gestation. Participants were part of the Maternal Adversity, Vulnerability, and Neurodevelopment (MAVAN) study, which examines the development of individual differences in phenotypes associated with multiple forms of psychopathology. Mothers were first assessed during their pregnancy (∼26 weeks) and then followed at multiple time points that included home visits and laboratory sessions.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Meaney, PhD, Study Director — James McGill Professor
Locations (1):
- Douglas Mental Health University Institute, Verdun, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Donnell KA, Gaudreau H, Colalillo S, Steiner M, Atkinson L, Moss E, Goldberg S, Karama S, Matthews SG, Lydon JE, Silveira PP, Wazana AD, Levitan RD, Sokolowski MB, Kennedy JL, Fleming A, Meaney MJ; MAVAN Research Team. The maternal adversity, vulnerability and neurodevelopment project: theory and methodology. Can J Psychiatry. 2014 Sep;59(9):497-508. doi: 10.1177/070674371405900906. PMID 25565695
- [Result] Mileva-Seitz V, Kennedy J, Atkinson L, Steiner M, Levitan R, Matthews SG, Meaney MJ, Sokolowski MB, Fleming AS. Serotonin transporter allelic variation in mothers predicts maternal sensitivity, behavior and attitudes toward 6-month-old infants. Genes Brain Behav. 2011 Apr;10(3):325-33. doi: 10.1111/j.1601-183X.2010.00671.x. Epub 2011 Jan 13. PMID 21232011
- [Result] Silveira PP, Agranonik M, Faras H, Portella AK, Meaney MJ, Levitan RD; Maternal Adversity, Vulnerability and Neurodevelopment Study Team. Preliminary evidence for an impulsivity-based thrifty eating phenotype. Pediatr Res. 2012 Mar;71(3):293-8. doi: 10.1038/pr.2011.39. Epub 2012 Jan 25. PMID 22278183
- [Result] Mileva-Seitz V, Steiner M, Atkinson L, Meaney MJ, Levitan R, Kennedy JL, Sokolowski MB, Fleming AS. Interaction between oxytocin genotypes and early experience predicts quality of mothering and postpartum mood. PLoS One. 2013 Apr 18;8(4):e61443. doi: 10.1371/journal.pone.0061443. Print 2013. PMID 23637833
- [Result] Jonas W, Mileva-Seitz V, Girard AW, Bisceglia R, Kennedy JL, Sokolowski M, Meaney MJ, Fleming AS, Steiner M; MAVAN Research Team. Genetic variation in oxytocin rs2740210 and early adversity associated with postpartum depression and breastfeeding duration. Genes Brain Behav. 2013 Oct;12(7):681-94. doi: 10.1111/gbb.12069. Epub 2013 Aug 31. PMID 23941164
- [Result] Adedinsewo DA, Fleming AS, Steiner M, Meaney MJ, Girard AW; MAVAN team. Maternal anxiety and breastfeeding: findings from the MAVAN (Maternal Adversity, Vulnerability and Neurodevelopment) Study. J Hum Lact. 2014 Feb;30(1):102-9. doi: 10.1177/0890334413504244. Epub 2013 Sep 24. PMID 24065719
- [Result] Silveira PP, Portella AK, Kennedy JL, Gaudreau H, Davis C, Steiner M, Soares CN, Matthews SG, Sokolowski MB, Dube L, Loucks EB, Hamilton J, Meaney MJ, Levitan RD; MAVAN Study Team. Association between the seven-repeat allele of the dopamine-4 receptor gene (DRD4) and spontaneous food intake in pre-school children. Appetite. 2014 Feb;73:15-22. doi: 10.1016/j.appet.2013.10.004. Epub 2013 Oct 20. PMID 24153108
- [Result] Neuwald MF, Agranonik M, Portella AK, Fleming A, Wazana A, Steiner M, Levitan RD, Meaney MJ, Silveira PP; MAVAN Study Team. Transgenerational effects of maternal care interact with fetal growth and influence attention skills at 18 months of age. Early Hum Dev. 2014 May;90(5):241-6. doi: 10.1016/j.earlhumdev.2014.01.015. Epub 2014 Mar 3. PMID 24602473
- [Result] Escobar RS, O'Donnell KA, Colalillo S, Pawlby S, Steiner M, Meaney MJ, Levitan RD, Silveira PP; MAVAN Study Team. Better quality of mother-child interaction at 4 years of age decreases emotional overeating in IUGR girls. Appetite. 2014 Oct;81:337-42. doi: 10.1016/j.appet.2014.06.107. Epub 2014 Jul 8. PMID 25014742
- [Result] Wendland BE, Atkinson L, Steiner M, Fleming AS, Pencharz P, Moss E, Gaudreau H, Silveira PP, Arenovich T, Matthews SG, Meaney MJ, Levitan RD; MAVAN Study Team. Low maternal sensitivity at 6 months of age predicts higher BMI in 48 month old girls but not boys. Appetite. 2014 Nov;82:97-102. doi: 10.1016/j.appet.2014.07.012. Epub 2014 Jul 15. PMID 25049136
- [Result] Pennestri MH, Moss E, O'Donnell K, Lecompte V, Bouvette-Turcot AA, Atkinson L, Minde K, Gruber R, Fleming AS, Meaney MJ, Gaudreau H; MAVAN Research Team. Establishment and consolidation of the sleep-wake cycle as a function of attachment pattern. Attach Hum Dev. 2015;17(1):23-42. doi: 10.1080/14616734.2014.953963. Epub 2014 Sep 18. PMID 25231054
- [Result] Levitan RD, Rivera J, Silveira PP, Steiner M, Gaudreau H, Hamilton J, Kennedy JL, Davis C, Dube L, Fellows L, Wazana A, Matthews S, Meaney MJ; MAVAN Study Team. Gender differences in the association between stop-signal reaction times, body mass indices and/or spontaneous food intake in pre-school children: an early model of compromised inhibitory control and obesity. Int J Obes (Lond). 2015 Apr;39(4):614-9. doi: 10.1038/ijo.2014.207. Epub 2014 Dec 16. PMID 25512364
- [Result] Bouvette-Turcot AA, Fleming AS, Wazana A, Sokolowski MB, Gaudreau H, Gonzalez A, Deslauriers J, Kennedy JL, Steiner M, Meaney MJ; MAVAN Research Team. Maternal childhood adversity and child temperament: an association moderated by child 5-HTTLPR genotype. Genes Brain Behav. 2015 Mar;14(3):229-37. doi: 10.1111/gbb.12205. Epub 2015 Mar 24. PMID 25688466
- [Result] Pennestri MH, Gaudreau H, Bouvette-Turcot AA, Moss E, Lecompte V, Atkinson L, Lydon J, Steiner M, Meaney MJ; Mavan Research Team. Attachment disorganization among children in Neonatal Intensive Care Unit: Preliminary results. Early Hum Dev. 2015 Oct;91(10):601-6. doi: 10.1016/j.earlhumdev.2015.07.005. Epub 2015 Aug 8. PMID 26261864
- [Result] Bouvette-Turcot AA, Pluess M, Bernier A, Pennestri MH, Levitan R, Sokolowski MB, Kennedy JL, Minde K, Steiner M, Pokhvisneva I, Meaney MJ, Gaudreau H; MAVAN research team. Effects of Genotype and Sleep on Temperament. Pediatrics. 2015 Oct;136(4):e914-21. doi: 10.1542/peds.2015-0080. Epub 2015 Sep 14. PMID 26371199
- [Result] Wazana A, Moss E, Jolicoeur-Martineau A, Graffi J, Tsabari G, Lecompte V, Pascuzzo K, Babineau V, Gordon-Green C, Mileva V, Atkinson L, Minde K, Bouvette-Turcot AA, Sassi R, St-Andre M, Carrey N, Matthews S, Sokolowski M, Lydon J, Gaudreau H, Steiner M, Kennedy JL, Fleming A, Levitan R, Meaney MJ. The interplay of birth weight, dopamine receptor D4 gene (DRD4), and early maternal care in the prediction of disorganized attachment at 36 months of age. Dev Psychopathol. 2015 Nov;27(4 Pt 1):1145-61. doi: 10.1017/S0954579415000735. PMID 26439067
- [Result] Reis RS, Bernardi JR, Steiner M, Meaney MJ, Levitan RD, Silveira PP; MAVAN Study Team. Poor infant inhibitory control predicts food fussiness in childhood - A possible protective role of n-3 PUFAs for vulnerable children. Prostaglandins Leukot Essent Fatty Acids. 2015 Jun;97:21-5. doi: 10.1016/j.plefa.2015.03.004. Epub 2015 Apr 3. PMID 25892188
- [Result] Babineau V, Green CG, Jolicoeur-Martineau A, Bouvette-Turcot AA, Minde K, Sassi R, St-Andre M, Carrey N, Atkinson L, Kennedy JL, Lydon J, Steiner M, Gaudreau H, Levitan R, Meaney M, Wazana A; MAVAN project. Prenatal depression and 5-HTTLPR interact to predict dysregulation from 3 to 36 months--a differential susceptibility model. J Child Psychol Psychiatry. 2015 Jan;56(1):21-9. doi: 10.1111/jcpp.12246. Epub 2014 May 15. PMID 24827922
- [Result] Silveira PP, Gaudreau H, Atkinson L, Fleming AS, Sokolowski MB, Steiner M, Kennedy JL, Meaney MJ, Levitan RD, Dube L. Genetic Differential Susceptibility to Socioeconomic Status and Childhood Obesogenic Behavior: Why Targeted Prevention May Be the Best Societal Investment. JAMA Pediatr. 2016 Apr;170(4):359-64. doi: 10.1001/jamapediatrics.2015.4253. PMID 26832777
- [Result] Cost KT, Plamondon A, Unternaehrer E, Meaney M, Steiner M, Fleming AS; MAVAN team. The more things change, the more things stay the same: maternal attitudes 3 to 18 months postpartum. Acta Paediatr. 2016 Jul;105(7):e320-7. doi: 10.1111/apa.13409. Epub 2016 May 6. PMID 26999290
- [Result] Green CG, Babineau V, Jolicoeur-Martineau A, Bouvette-Turcot AA, Minde K, Sassi R, St-Andre M, Carrey N, Atkinson L, Kennedy JL, Steiner M, Lydon J, Gaudreau H, Burack JA, Levitan R, Meaney MJ, Wazana A; Maternal Adversity, Vulnerability, and Neurodevelopment Research Team. Prenatal maternal depression and child serotonin transporter linked polymorphic region (5-HTTLPR) and dopamine receptor D4 (DRD4) genotype predict negative emotionality from 3 to 36 months. Dev Psychopathol. 2017 Aug;29(3):901-917. doi: 10.1017/S0954579416000560. Epub 2016 Jul 18. PMID 27427178
- [Result] Bouvette-Turcot AA, Unternaehrer E, Gaudreau H, Lydon JE, Steiner M, Meaney MJ; MAVAN Research Team. The joint contribution of maternal history of early adversity and adulthood depression to socioeconomic status and potential relevance for offspring development. J Affect Disord. 2017 Jan 1;207:26-31. doi: 10.1016/j.jad.2016.08.012. Epub 2016 Aug 16. PMID 27685851
- [Result] Tombeau Cost K, Unternaehrer E, Plamondon A, Steiner M, Meaney M, Atkinson L, Kennedy JL, Fleming AS; MAVAN Research Team. Thinking and doing: the effects of dopamine and oxytocin genes and executive function on mothering behaviours. Genes Brain Behav. 2017 Feb;16(2):285-295. doi: 10.1111/gbb.12337. Epub 2016 Oct 21. PMID 27620964
- [Result] Levitan RD, Jansen P, Wendland B, Tiemeier H, Jaddoe VW, Silveira PP, Kennedy JL, Atkinson L, Fleming A, Sokolowski M, Gaudreau H, Steiner M, Dube L, Hamilton J, Moss E, Wazana A, Meaney M. A DRD4 gene by maternal sensitivity interaction predicts risk for overweight or obesity in two independent cohorts of preschool children. J Child Psychol Psychiatry. 2017 Feb;58(2):180-188. doi: 10.1111/jcpp.12646. Epub 2016 Oct 11. PMID 27726127
- [Result] Maunder RG, Hunter JJ, Atkinson L, Steiner M, Wazana A, Fleming AS, Moss E, Gaudreau H, Meaney MJ, Levitan RD. An Attachment-Based Model of the Relationship Between Childhood Adversity and Somatization in Children and Adults. Psychosom Med. 2017 Jun;79(5):506-513. doi: 10.1097/PSY.0000000000000437. PMID 27941580
- [Result] Pokhvisneva I, Leger E, Meaney MJ, Silveira PP. Systematic Overestimation of Reflection Impulsivity in the Information Sampling Task: Age Dependency in Children. Biol Psychiatry. 2018 Jan 15;83(2):e33-e34. doi: 10.1016/j.biopsych.2016.12.027. Epub 2017 Jan 5. No abstract available. PMID 28189253
- [Result] Bischoff AR, Pokhvisneva I, Leger E, Gaudreau H, Steiner M, Kennedy JL, O'Donnell KJ, Diorio J, Meaney MJ, Silveira PP; MAVAN research team. Dynamic interaction between fetal adversity and a genetic score reflecting dopamine function on developmental outcomes at 36 months. PLoS One. 2017 May 15;12(5):e0177344. doi: 10.1371/journal.pone.0177344. eCollection 2017. PMID 28505190
- [Result] Silveira PP, Pokhvisneva I, Gaudreau H, Atkinson L, Fleming AS, Sokolowski MB, Steiner M, Kennedy JL, Dube L, Levitan RD, Meaney MJ; MAVAN research team. Fetal growth interacts with multilocus genetic score reflecting dopamine signaling capacity to predict spontaneous sugar intake in children. Appetite. 2018 Jan 1;120:596-601. doi: 10.1016/j.appet.2017.10.021. Epub 2017 Oct 14. PMID 29038017
- [Result] Graffi J, Moss E, Jolicoeur-Martineau A, Moss G, Lecompte V, Pascuzzo K, Babineau V, Gordon-Green C, Mileva-Seitz VR, Minde K, Sassi R, Steiner M, Kennedy JL, Gaudreau H, Levitan R, Meaney MJ, Wazana A; MAVAN project. The dopamine D4 receptor gene, birth weight, maternal depression, maternal attention, and the prediction of disorganized attachment at 36 months of age: A prospective genexenvironment analysis. Infant Behav Dev. 2018 Feb;50:64-77. doi: 10.1016/j.infbeh.2017.11.004. Epub 2017 Nov 21. PMID 29149620
- [Result] Parent C, Pokhvisneva I, Gaudreau H, Diorio J, Meaney MJ, Silveira PP; MAVAN Research Team. Community study found that cutaneous allergies in childhood were associated with conduct problems in girls. Acta Paediatr. 2018 May;107(5):900-901. doi: 10.1111/apa.14235. Epub 2018 Feb 19. No abstract available. PMID 29364555
- [Result] Silveira PP, Pokhvisneva I, Gaudreau H, Rifkin-Graboi A, Broekman BFP, Steiner M, Levitan R, Parent C, Diorio J, Meaney MJ. Birth weight and catch up growth are associated with childhood impulsivity in two independent cohorts. Sci Rep. 2018 Sep 12;8(1):13705. doi: 10.1038/s41598-018-31816-5. PMID 30209275
- [Result] Jolicoeur-Martineau A, Wazana A, Szekely E, Steiner M, Fleming AS, Kennedy JL, Meaney MJ, Greenwood CMT. Alternating optimization for G x E modelling with weighted genetic and environmental scores: Examples from the MAVAN study. Psychol Methods. 2019 Apr;24(2):196-216. doi: 10.1037/met0000175. Epub 2018 Aug 13. PMID 30102054
- [Result] Belsky J, Pokhvisneva I, Rema ASS, Broekman BFP, Pluess M, O'Donnell KJ, Meaney MJ, Silveira PP. Polygenic differential susceptibility to prenatal adversity. Dev Psychopathol. 2019 May;31(2):439-441. doi: 10.1017/S0954579418000378. Epub 2018 Aug 7. PMID 30081968
- [Result] Laganiere C, Gaudreau H, Pokhvisneva I, Atkinson L, Meaney M, Pennestri MH. Maternal characteristics and behavioural/emotional problems in preschoolers: how they relate to sleep rhythmic movements at sleep onset. J Sleep Res. 2019 Jun;28(3):e12707. doi: 10.1111/jsr.12707. Epub 2018 Jun 5. PMID 29873138
- [Result] Garg E, Chen L, Nguyen TTT, Pokhvisneva I, Chen LM, Unternaehrer E, MacIsaac JL, McEwen LM, Mah SM, Gaudreau H, Levitan R, Moss E, Sokolowski MB, Kennedy JL, Steiner MS, Meaney MJ, Holbrook JD, Silveira PP, Karnani N, Kobor MS, O'Donnell KJ; Mavan Study Team. The early care environment and DNA methylome variation in childhood. Dev Psychopathol. 2018 Aug;30(3):891-903. doi: 10.1017/S0954579418000627. PMID 30068421
- [Result] Jonas W, Bisceglia R, Meaney MJ, Dudin A, Fleming AS, Steiner M; MAVAN Research Team. The role of breastfeeding in the association between maternal and infant cortisol attunement in the first postpartum year. Acta Paediatr. 2018 Jul;107(7):1205-1217. doi: 10.1111/apa.14256. Epub 2018 Mar 24. PMID 29405436
- [Result] Forest M, O'Donnell KJ, Voisin G, Gaudreau H, MacIsaac JL, McEwen LM, Silveira PP, Steiner M, Kobor MS, Meaney MJ, Greenwood CMT. Agreement in DNA methylation levels from the Illumina 450K array across batches, tissues, and time. Epigenetics. 2018;13(1):19-32. doi: 10.1080/15592294.2017.1411443. Epub 2018 Jan 30. PMID 29381404
- [Result] Silveira PP, Pokhvisneva I, Parent C, Cai S, Rema ASS, Broekman BFP, Rifkin-Graboi A, Pluess M, O'Donnell KJ, Meaney MJ. Cumulative prenatal exposure to adversity reveals associations with a broad range of neurodevelopmental outcomes that are moderated by a novel, biologically informed polygenetic score based on the serotonin transporter solute carrier family C6, member 4 (SLC6A4) gene expression. Dev Psychopathol. 2017 Dec;29(5):1601-1617. doi: 10.1017/S0954579417001262. PMID 29162172
- [Result] Agranonik M, Portella AK, Hamilton J, Fleming AS, Steiner M, Meaney MJ, Levitan RD, Silveira PP; MAVAN study team. Breastfeeding in the 21st century. Lancet. 2016 May 21;387(10033):2088-2089. doi: 10.1016/S0140-6736(16)30536-0. No abstract available. PMID 27301818
- [Result] Jonas W, Atkinson L, Steiner M, Meaney MJ, Wazana A, Fleming AS; MAVAN research team. Breastfeeding and maternal sensitivity predict early infant temperament. Acta Paediatr. 2015 Jul;104(7):678-86. doi: 10.1111/apa.12987. Epub 2015 Apr 22. PMID 25727570
- [Result] Graffi J, Moss E, Jolicoeur-Martineau A, Moss G, Lecompte V, Pascuzzo K, Babineau V, Gordon-Green C, Mileva-Seitz VR, Minde K, Sassi R, Carrey N, Kennedy JL, Gaudreau H, Levitan R, Meaney M, Wazana A. Preschool children without 7-repeat DRD4 gene more likely to develop disorganized attachment style. McGill Sci Undergrad Res J. 2015 Mar;10(1):31-36. PMID 28574063
- [Result] Agrati D, Browne D, Jonas W, Meaney M, Atkinson L, Steiner M, Fleming AS; MAVAN research team. Maternal anxiety from pregnancy to 2 years postpartum: transactional patterns of maternal early adversity and child temperament. Arch Womens Ment Health. 2015 Oct;18(5):693-705. doi: 10.1007/s00737-014-0491-y. Epub 2015 Jan 29. PMID 25627018
- [Result] Plamondon A, Akbari E, Atkinson L, Steiner M, Meaney MJ, Fleming AS; MAVAN research team. Spatial working memory and attention skills are predicted by maternal stress during pregnancy. Early Hum Dev. 2015 Jan;91(1):23-9. doi: 10.1016/j.earlhumdev.2014.11.004. Epub 2014 Nov 26. PMID 25460253

RESULTS

PARTICIPANT FLOW:
Groups:
- Prenatal and 3 to 72 Months: Our community sample consisted of mothers recruited in Montréal (Québec) and Hamilton (Ontario), Canada, at 13 to 20 weeks' gestation. Participants were part of the Maternal Adversity, Vulnerability, and Neurodevelopment (MAVAN) study, which examines the development of individual differences in phenotypes associated with multiple forms of psychopathology. Mothers were first assessed during their pregnancy (∼26 weeks) and then followed at multiple time points that included home visits and laboratory sessions.
Period: Overall Study
Arm/Group | Prenatal and 3 to 72 Months
Started | 630
Completed | 630
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 630
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 288
  Male | 342
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of Participants that Provided Feedback on the Childhood Trauma Questionnaire [Count of Participants; unit: Participants] | 429

OUTCOME MEASURES:

1. Primary Outcome: Child's Cognitive Development Measured Using the Bayley Scales of Infant Development II.
Description: Assessment of child development was done using the cognitive, motor and mental scales of the Bayley Scales of Infant Development II.
Time Frame: At 6, 12, 18 and 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  6 months | 524
  12 months | 508
  18 months | 458
  36 months | 422

2. Primary Outcome: Child Temperament Evaluated Using the Infant Behaviour Questionnaire.
Description: Child temperament was evaluated using the Infant Behaviour questionnaire (IBQ). The items represent 14 scales but factor analysis reveals three primary factors: a) impulsivity, b) negative affectivity and c) effortful control.
Time Frame: 3 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  3 months | 387
  6 months | 475

3. Primary Outcome: Changes in Child Temperament Evaluated Using the Early Childhood Behaviour Questionnaire.
Description: Assessment of child's temperament was done with the Early Childhood Behaviour questionnaire, the toddler version of the IBQ. It is comprised of 201 items grouped in 18 subscales and is based on a 7-point Likert scale ranging from "never" to "always". The questionnaire yields 18 sub-scores: activity level/energy, attentional focusing, attentional shifting, cuddliness, fear, frustration, high-intensity pleasure, impulsivity, inhibitory control, low-intensity pleasure, motor activation, perceptual sensitivity, positive anticipation, sadness, shyness, sociability, and soothability.
Time Frame: 18 and 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  18 months | 433
  36 months | 420

4. Primary Outcome: Changes in Socio-emotional Development Measured Using the Infant Toddler Socio-emotional Assessment Questionnaire.
Description: Socio-emotional development was measured using the Infant Toddler Socio-emotional Assessment questionnaire (ITSEA). It consists of 140 items to evaluate four independent behavioral domains: 1) externalizing, (e.g., high-activity, aggression, defiance, and negative emotional reactivity); 2) internalizing, (e.g., mood regulation problems, social withdrawal and extreme inhibition/shyness); 3) dysregulation (e.g., sleep and eating problems, mood regulation); and 4) maladaptation (e.g., repetitive and stereotypic behaviors). Items are rated on a 3-point scale.
Time Frame: 18 and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  18 months | 485
  24 months | 471

5. Primary Outcome: Changes in Child's Behaviour Problems Measured With the Child Behaviour Checklist.
Description: Child's behaviour was evaluated using the Child Behaviour Checklist (CBCL). The CBCL is a well-validated screen for childhood psychopathology. This parent-rated questionnaire contains 100 items divided in 2 broad scales :
  Internalizing problems includes : Withdrawn, Somatic Complaints, and Anxious/Depressed subscales. Externalizing problems : including Rule-Breaking Behavior and Aggressive subscales. Total problems score : is the sum of the scores of all the problem items.
Time Frame: 48 and 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  48 months | 366
  60 months | 310

6. Primary Outcome: Changes in Child's School Readiness Measured With the School Readiness Test Battery.
Description: School and academic readiness were assessed using the School readiness test battery, including the Lollipop test, Number knowledge and Peabody Picture Vocabulary test.
  The NKT measures the development of number concepts. This test measures the mastery of a series of concepts required for learning math and comprises 5 levels.
  The Lollipop includes 52 questions, divided in 4 knowledge subtests: (1) colours and forms, (2) spatial relationships, (3) numbers and (4) letters. It is a good predictor of reading and math achievement up to 4th grade.
  The PPVT is a receptive vocabulary test that measures the extent of vocabulary a child can understand. A child is asked to identify a spoken word on an array of four pictures, only one of which is correct.
Time Frame: 48 and 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  48 months | 366
  60 months | 322

7. Primary Outcome: Evaluation or Child's Cognitive Development Using the Developmental Neuropsychological Assessment.
Description: Child's cognitive development was assessed using the sensory-motor and visuo-spatial processing subscales of the Developmental Neuropsychological Assessment (NEPSY).
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 358

8. Primary Outcome: Evaluation of Child's Cognitive Development Using the Weschler Preschool and Primary Scale of Intelligence.
Description: Child's cognitive development was assessed using the vocabulary and the bloc design subscales of the Weschler Preschool Primary Scale of Intelligence (WPPSI).
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 355

9. Primary Outcome: Changes in Child's Hyperactivity Problems Measured With the Conner's.
Description: The Conner's was designed to be completed by parents and teachers to assist in evaluating children for attention-deficit/hyperactivity disorder (ADHD). The parents' short version contains 27 items and the teachers' short version has 28. The teacher version is similar but lacks the psychosomatic scale contained on the parent version. The Conner's is validated and the standard for informant-administered ADHD assessment both in clinical and research settings. Oppositional, cognitive problems/inattention, hyperactivity subscales.
Time Frame: 60 and 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  60 months | 323
  72 months | 272

10. Primary Outcome: Child's Fears Assessed With the Koala Fear Questionnaire.
Description: The Koala Fear Questionnaire (KFQ) is a standardized self-report scale for assessing fears and fearfulness in children aged between 4 and 12 years. This scale consists of 31 potentially fear-provoking stimuli and situations that are all illustrated with pictures. Children rate the intensity of their fear of these stimuli by using a visual scale depicting Koala bears expressing various degrees of fear ( no fear, some fear, a lot of fear ).
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 353

11. Primary Outcome: Changes in Child's Emotional and Behaviour Problems Measured With the Strength and Difficulty Questionnaire.
Description: The Strengths and Difficulties Questionnaire (SDQ) is a brief screening for child emotional and behavioural problems.
  It is based on 25 items on psychological attributes.
  1. emotional symptoms (5 items)
  2. conduct problems (5 items)
  3. hyperactivity/inattention (5 items)
  4. peer relationship problems (5 items)
  5. prosocial behaviour (5 items) Number 1) to 4) added together to generate a total difficulties score.
Time Frame: 60 and 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  60 months | 323
  72 months | 271

12. Primary Outcome: Child's Behavioural Inhibition and Behavioural Activation Were Measured Using the Behavioural Inhibition System (BIS) and the Behavioural Approach System (BAS)
Description: The BIS/BAS was designed to assess dispositional sensitivity to the behavioral inhibition system (BIS) and the behavioral activation or behavioral approach system (BAS).
  Questions 20 items using 4 point scales (1 = strongly disagree to 4 = strongly agree).
  2 subscales: Behavioral Inhibition System (BIS) 7 items about anticipation of punishment Behavioral Action System (BAS), which has 3 subscales of its own: Reward Responsiveness (RR) 5 items about anticipation or occurrence of reward Drive (D) 4 items about pursuit of desired goals. Fun Seeking (FS) 4 items about desire for new rewards and impulsive approach to potential rewards.
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 303

13. Primary Outcome: Child's Mental Health Was Evaluated Using the Dominic Questionnaire.
Description: The Dominic questionnaire is a structured pictorial instrument assessing mental disorders in 6- to 11-year-old children. The Dominic assesses a child's perception of her/his own symptoms, which is critical to balance parents' and school professionals' perception. Ninety-nine drawings represent situations corresponding to DSM-III-R based. ADHD, Conduct Disorder, Oppositional Defiant Disorder, Major Depressive Disorder, Separation Anxiety Disorder, Generalized Anxiety Disorder and Specific Phobia.
Time Frame: 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 279

14. Primary Outcome: The Child's Attributional Style Was Evaluated With the Child Attributional Style Interview.
Description: The Child Attributional Style Interview (CASI) is a measure of attributional style in children aged five years old and older. The interactive interview consists of sixteen events, which are presented to the child as illustrations, in a storybook format. The events are equally divided on two domains: valence (positive and negative theme), and interpersonal (parents and peers) and achievement. This creates the possibility of four sub-categories for analysis (i.e. positive-achievement, negative-interpersonal etc.). After the presentation of each event, the child is asked three questions for their level of internal, stable and global attributions for each event.
Time Frame: 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 275

15. Primary Outcome: Changes in Child's Feeding Behaviour Was Measured With the Child Eating Behaviour Questionnaire.
Description: The Child Eating Behaviour Questionnaire (CEBQ) was designed to assess children's eating scale styles. It is a parent-report measure comprised of 35 items, each rated on a five-point likert scale that ranges from never to always. The instrument is ideal for use in research investigating the early precursors of eating disorders or obesity.
Time Frame: 48 and 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  48 months | 395
  72 months | 305

16. Primary Outcome: Child's Executive Functioning Measured With the Behavior Rating of Executive Function.
Description: The Behavior Rating Inventory of Executive Function (BRIEF) measures executive function behaviors for children and adolescents ages 5-18. Each form of the BRIEF parent- and teacher- rating form contains 86 items in eight non-overlapping clinical scales and two validity scales. These theoretically and statistically derived scales form two indexes: a) Behavioral Regulation (three scales) and b) Metacognition (five scales), as well as a Global Executive Composite score which takes into account all of the clinical scales and represents the child's overall executive function.
Time Frame: 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 307

17. Primary Outcome: Sensitivity to Punishment & Sensitivity to Reward in Children Will be Evaluated Using the Child Version of the Sensitivity to Punishment & Sensitivity to Reward Questionnaire.
Description: The Sensitivity to Punishment & Sensitivity to Reward questionnaire (SPSRQ-C) measures parent-rated sensitivity to punishment and reward and contains 33 items, divided in a Punishment Sensitivity scale, and three Reward Sensitivity scales: Reward Responsivity, Impulsivity/Fun-Seeking, and Drive. Each item is scored on a 5-point Likert scale.
Time Frame: 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 308

18. Secondary Outcome: Changes in Mother's Depression Symptoms Measured With the Beck Depression Inventory.
Description: The Beck Depression Inventory (BDI-II) is a 21-question multiple-choice self-report inventory that is one of the most widely used instruments for measuring the severity of depression. The most current version of the questionnaire is designed for individuals aged 13 and over and is composed of items relating to depression symptoms such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex (15 minutes). BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63.
Time Frame: 60 and 72 months
Population: The data is currently being analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  60 months | 318
  72 months | 261

19. Secondary Outcome: Changes in Mother's Depression Symptoms Measured With the Center for Epidemiological Studies, Depression Scale.
Description: The Center for Epidemiological Studies, Depression Scale (CES-D) is a 20-item instrument that has excellent internal consistency (.90) and reasonable test-retest reliability (.54) for a scale that should be sensitive to adverse changes in the respondent's environment. Questions ake to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Time Frame: Prenatal, 6, 12, 24, 36, 48, 60, 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  prenatal | 533
  6 months | 554
  12 months | 518
  24 months | 471
  36 months | 437
  48 months | 391
  60 months | 342
  72 months | 287

20. Secondary Outcome: Changes in Mother's Depression Symptoms Were Measured With the Edinburgh Postnatal Depression Scale.
Description: Edinburgh Postnatal Depression Scale (EPDS). The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report scale designed to screen for postpartum depression. The scale consists of 10 short statements with four possible answers corresponding to how the mother has felt during the past week. Responses are scored 0, 1, 2 and 3 based on the seriousness of the symptom. A higher total sum score indicates more severe symptoms of depression.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 481

21. Secondary Outcome: Changes in Mother's Anxiety Symptoms Were Measured Using the Speilberger State-Trait Anxiety Inventory.
Description: The Speilberger State-Trait Anxiety Inventory (STAI) is self-report scale consisting of two forms of 20 items each to measure psychic components of state and trait anxiety. The State-Anxiety scale measures intensity of current feelings "at this moment": 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. The Trait-Anxiety scale measures the frequency of feelings "in general": 1) almost never, 2) sometimes, 3) often, and 4) almost always.
Time Frame: 3, 24 and 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants
  3 months | 410
  24 months | 471
  60 months | 338

22. Secondary Outcome: Mother's Retrospective Assessment of Parental Educational Style Using the Parental Bonding Inventory.
Description: Parental Bonding Inventory (PBI) is a standard in retrospective assessment of parental educational style (48 items). Two scales termed 'care' and 'overprotection' or 'control', measure fundamental parental styles as perceived by the child. The measure is 'retrospective', meaning that adults (over 16 years) complete the measure for how they remember their parents during their first 16 years. The measure is to be completed for both mothers and fathers separately. There are 25 item questions, including 12 'care' items and 13 'overprotection' items.
Time Frame: 6 months
Population: The data is currently being analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 475

23. Secondary Outcome: Changes in Mother's Sensitivity Was Evaluated Using the Maternal Behaviour Q Sort (Short Version) and the Ainsworth Scales.
Description: Mother's sensitivity was assessed using the Maternal Behaviour Q sort (short version) and the Ainsworth scales (AINS). MBQS-S and AINS assess maternal sensitivity. Trained raters scored the mother's behavior on the scale for the MBQS and four scales of the AINS scales (Acceptance, Availability, Cooperation and Sensitivity) during a 20 and 30 minutes video-taped home mother-child interaction. The scales range from -1 to 1 for the MBQS and from 1 to 9 for the AINS scales, with higher scores indicating highly sensitive mothers on both instruments.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 99

24. Secondary Outcome: Mother's Early Life Abuse and Neglect Were Evaluated Using the Childhood Trauma Questionnaire.
Description: The Childhood Trauma Questionnaire (CTQ) is a 28-item self-report retrospective inventory intending to measure childhood or adolescent abuse and neglect, on a 5-point Likert scale ranging from Never True to Very Often True. The central constructs underlying the questionnaire are emotional, physical neglect and abuse, and sexual abuse. The CTQ contains five subscales :
  3 subscales assessing abuse : Emotional, Physical, and Sexual abuse 2 subscales assessing neglect : Emotional and Physical neglect.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 429

25. Secondary Outcome: Mother's Eating Behaviours Were Evaluated Using the Dutch Eating Behavior Questionnaire.
Description: The Dutch Eating Behavior Questionnaire is used to assess emotional, external and restrained eating. The 33 items on the DEBQ represent three separate scales: (i) Emotional Eating, with items such as 'Do you have the desire to eat when you are irritated?, contains 13 items; (ii) External Eating, with items such as 'Do you eat more than usual when you see others eating?, includes 10 items; and (iii) Restraint, with items such as 'Do you deliberately eat less in order not to become heavier? ', has 10 items.
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 350

26. Secondary Outcome: Mother's Sensitivity to Punishment and Sensitivity to Reward Were Measured Using the Sensitivity to Punishment and Sensitivity to Reward Questionnaire.
Description: The Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ) (Torrubia et al., 2001) is a 48 yes/no questionnaire measuring SP (sensitivity to punishment) and SR (sensitivity to reward) functioning.
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 350

27. Secondary Outcome: Parenting Style Assessed Using the Parental Authority Questionnaire.
Description: The Parental Authority Questionnaire (PAQ) investigates three prototypes of parental behavior: permissive, authoritative and authoritarian. Each prototype is measured on 10 items on a Likert scale from 1 (disagree strongly) to 5 (agree strongly). The questionnaire was developed to be answered by the child, however, it was adapted in order to let the mother rate her own prototype of parenting. Item scores for each scale were averaged to obtain a total prototype score, with high scores indicating that the mother rates herself to engage strongly in a given parenting prototype.
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 323

28. Secondary Outcome: Family Functioning Assessed Using the Family Assessment Device Questionnaire.
Description: The Family Assessment Device (FAD) questionnaire assesses family functioning on each dimension of the McMaster Model of Family Functioning (MMFF) according to individual family member's perception of their family's functioning. In addition to the six subscales of the MMFF (Problem solving, communication, roles, affective responsiveness, affective involvement, behaviour control) the FAD includes a General Functioning scale that measures the overall level of the family's functioning. Sixty statements, geared to an eighth-grade reading level, describe various aspects of family functioning. Each member of the family over the age of 12 completes the pen-and-paper questionnaire by rating how well the statement describes his or her family. There are four choices (strongly agree, agree, disagree, strongly disagree) per item for each dimension. Dimension items are purposely not listed in consecutive order. Each item matches only one dimension and may describe healthy or unhealthy functioning.
Time Frame: 72 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal and 3 to 72 Months
Number analyzed (Participants) | 630
Participants | 307

ADVERSE EVENTS:
Time Frame: 6 years
Description: The study is observational and not experimental. No adverse events were unforeseen for data collection tools used in the study.
Groups:
- Adverse Events: all adverse events
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/630
Serious Adverse Events (participants affected / at risk) | 0/630
Other Adverse Events (participants affected / at risk) | 0/630

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Original cohort prenatal-48 months (2004-02-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03434457/Prot_SAP_000.pdf
  • Study Protocol: 60 months amendment (2008-06-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03434457/Prot_001.pdf
  • Study Protocol: 72 months amendment (2009-10-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT03434457/Prot_002.pdf